CLINICAL TRIAL: NCT00989508
Title: Myocardial Protection With Perhexiline in Left Ventricular Hypertrophy
Acronym: HYPER
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: University of Birmingham (Other); Brighton and Sussex University Hospitals NHS Trust (Other); British Heart Foundation (Other)
Responsible Party: Mr Domenico Pagano, University Hospital Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRK3535; Eudract 2008-002376-95; REC 08/H0304/48; BHF PG/08/040
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-04

CONDITIONS: Myocardial Reperfusion Injury; Cardiac Output, Low; Hypertrophy, Left Ventricular
Keywords: Perhexiline; Aortic Valve Stenosis; Hypertrophy, Left Ventricular; Myocardial Reperfusion Injury; Cardiac Output, Low; Troponin
MeSH Terms: conditions — Myocardial Reperfusion Injury; Cardiac Output, Low; Hypertrophy, Left Ventricular; Aortic Valve Stenosis | interventions — Perhexiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perhexiline (Experimental): Pre-operative administration of Perhexiline tablets according to dosing schedule
  Interventions: Drug: Perhexiline
- Placebo marked PEXSIG (Placebo Comparator): Pre-operative administration of placebo tablets according to dosing schedule
  Interventions: Drug: Placebo marked PEXSIG

INTERVENTIONS:
Drug: Perhexiline — Tablets. Dose: 200mg BD for 3 days, then 100mg BD until surgery. Duration of therapy: 5-31 days.
  Other Names: PEXSIG
  Arms: Perhexiline
Drug: Placebo marked PEXSIG — Tablets. Dose: 200mg BD for 3 days, then 100mg BD until surgery. Duration of therapy: 5-31 days.
  Arms: Placebo marked PEXSIG

SUMMARY:
Open-heart surgery causes injury of the heart muscle. Although this is usually mild, temporary and reversible, if it is severe it can endanger life and require additional high cost care. During surgery, techniques are used to protect the heart from injury, but these remain imperfect. Patients with a thickened wall of the heart (left ventricular hypertrophy) may be at greater risk. This study assesses the effect of facilitating sugar metabolism (a more efficient fuel) by the heart muscle using the drug Perhexiline given before the operation.

This treatment has a sound experimental basis for improving outcome. If this improvement is confirmed surgical results could be improved. The investigators will be studying heart function, heart muscle energy stores and chemicals which quantify the amount of heart muscle injury. The investigators' hypothesis is that Perhexiline will improve the protection of the heart by decreasing damage that may occur during heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* First-time
* Aortic valve surgery for aortic stenosis +/- coronary artery bypass

Exclusion Criteria:

* Diabetes Mellitus
* Renal impairment with Creatinine greater than or equal to 200micromol/L
* Atrial fibrillation
* Amiodarone therapy, recent (in last month) or current
* Hepatic impairment, significant preoperative
* Peripheral neuropathy
* Pregnancy or breast-feeding
* Emergency surgery or required on clinical grounds within 5 days of referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Absolute difference in Cardiac Index (>0.3 l/min/m2) | 6 hours post-removal of aortic X-clamp

SECONDARY OUTCOMES:
Incidence of Low Cardiac Output Syndrome | 6 hours post-removal of aortic X-clamp
Incidence of inotrope use according to protocol | 6 and 12 hours post-removal of aortic X-clamp
Peak and total release of Troponin | 12 and 24 hours post-release of aortic X-clamp

CONTACTS AND LOCATIONS:
Overall Officials: Domeinco Pagano, MD FRCS, Principal Investigator — University Hospital Birmingham
Locations (1):
- University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Quinn DW, Pagano D, Bonser RS, Rooney SJ, Graham TR, Wilson IC, Keogh BE, Townend JN, Lewis ME, Nightingale P; Study Investigators. Improved myocardial protection during coronary artery surgery with glucose-insulin-potassium: a randomized controlled trial. J Thorac Cardiovasc Surg. 2006 Jan;131(1):34-42. doi: 10.1016/j.jtcvs.2005.05.057. PMID 16399292
- [Background] Ranasinghe AM, Quinn DW, Pagano D, Edwards N, Faroqui M, Graham TR, Keogh BE, Mascaro J, Riddington DW, Rooney SJ, Townend JN, Wilson IC, Bonser RS. Glucose-insulin-potassium and tri-iodothyronine individually improve hemodynamic performance and are associated with reduced troponin I release after on-pump coronary artery bypass grafting. Circulation. 2006 Jul 4;114(1 Suppl):I245-50. doi: 10.1161/CIRCULATIONAHA.105.000786. PMID 16820580
- [Background] Ashrafian H, Horowitz JD, Frenneaux MP. Perhexiline. Cardiovasc Drug Rev. 2007 Spring;25(1):76-97. doi: 10.1111/j.1527-3466.2007.00006.x. PMID 17445089